CLINICAL TRIAL: NCT06675773
Title: The Effect of Conscious Awareness Development Psychoeducation Program Prepared for Caregivers on Conscious Awareness, Job Stress and Compassion Fatigue.
Brief Title: The Effect of Conscious Awareness Development Psychoeducation Program Prepared for Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Nilüfer KIRANŞAL, Lecturer, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KAÜ-SBF-NK 01
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Mental Health Issue
Keywords: Mindfulness,; Work stress; Compassion Fatigue; Psychoeducation
MeSH Terms: conditions — Occupational Stress; Compassion Fatigue

STUDY DESIGN:
Intervention Model Description: Two groups were mindfulness-based psychoeducation controls.
Who Masked: Investigator
Masking Description: The training will be conducted by the investigator. The experimental and control groups will be assigned by a statistics expert other than the investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The Conscious Awareness Development Psychoeducation Program will be applied to the experimental group. Conscious awareness and self-compassion techniques will be used in the psychoeducation program sessions. Homework will be given to the participants in each session. The psychoeducation program is prepared based on conscious awareness.
  Interventions: Other: Conscious Awareness Development Psychoeducation Program
- Control Group (No Intervention): No application will be made to the Control Group.

INTERVENTIONS:
Other: Conscious Awareness Development Psychoeducation Program — The Conscious Awareness Development Psychoeducation Program consists of nine sessions. The sessions will be applied once a week and last 90 minutes. The psychoeducation program is prepared based on conscious awareness. Conscious awareness and self-compassion techniques will be used in the sessions. Homework will be given to the participants in each session.
  Arms: Experimental Group

SUMMARY:
This study aimed to increase the conscious awareness of caregivers and reduce work stress and compassion fatigue.

DETAILED DESCRIPTION:
This study was planned in an experimental design with pre-test post-test follow-up measurements, experimental and control groups. The universe of the study consisted of care personnel working in institutions affiliated to the Provincial Directorate of Family, Labor and Social Services located in a city center in the east of Turkey. The sample calculation was made using the G-Power program (Experiment 14, Control 14). Since there may be omissions, the experimental group was determined as 20 participants and the control group as 20 participants. In this study, a nine-session training program will be applied to the experimental group. No application will be made to the control group. The conscious awareness development psychoeducation program will be applied once a week and for 90 minutes. Each session will be conducted in line with certain objectives. The sessions will be conducted by the investigator. Ethics committee approval was obtained before starting the study. Institutional permissions and written informed consent will be obtained for the participants. Informed consent will include information about the research and information that will ensure confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Being actively working as a care worker in relevant institutions.

Exclusion Criteria:

* Having received similar training before
* Having been diagnosed with a mental illness
* Wanting to leave the study at any stage.
* Not having attended more than two sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
The Mindful Attention Awareness Scale-MAAS | Pre-test -Post-test (9 weeks) Follow-up ( 3 month after)
  Originally named The Mindful Attention Awareness Scale-MAAS, it measures the attention and present time awareness of an individual in their daily lives. It consists of 15 items and a single sub-dimension. The scale is in the form of a 6-point Likert and is evaluated as a single total score. Individuals who score high on the scale show that their conscious awareness levels are high (Brown and Rayn 2003, Özyeşil et al. 2011)

SECONDARY OUTCOMES:
General Work Stress Scale | Pre-test -Post-test (9 weeks) Follow-up ( 3 month after)
  The General Job Stress Scale evaluates the level of stress that an individual experiences or perceives in relation to work in general. The scale, which consists of 9 items and a single dimension, is in the form of a 5-point Likert. High scores on the scale indicate high job stress, and low scores indicate low job stress (Teleş 2021).
Compassion Fatigue Scale- Short Scale Form | Pre-test -Post-test (9 weeks) Follow-up ( 3 month after)
  The scale consists of 13 items and two sub-dimensions: secondary trauma and occupational burnout. The lowest score possible from the 10-point Likert-type scale is 13 and the highest is 130. As the scores increase, the level of compassion fatigue experienced by individuals also increases (Dinç and Ekinci, 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer KIRANŞAL, Principal Investigator — Lecturer
Locations (1):
- Faculty of Health Sciences Kafkas University, Kars, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: the General Work Stress Scale — https://toad.halileksi.net/wp-content/uploads/2022/07/genel-is-stresi-olcegi-toad.pdf
- See also: Compassion Fatigue Short Scale — https://dergipark.org.tr/en/pub/pgy/article/590616